CLINICAL TRIAL: NCT01520519
Title: A Phase 2 Study of the Combination of the Bruton's Tyrosine Kinase Inhibitor PCI-32765 and Rituximab in High-Risk Chronic Lymphocytic Leukemia (CLL) and Small Lymphocytic Lymphoma (SLL) Patients
Brief Title: Phase 2 Study of the Combination of Bruton's Tyrosine Kinase Inhibitor PCI-32765 and Rituximab in High-Risk Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0785; NCI-2012-00126 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Results first posted 2019-09-18 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Leukemia
Keywords: Leukemia; Chronic Lymphocytic Leukemia; CLL; Small Lymphocytic Lymphoma; SLL; Rituximab; Rituxan; PCI-32765
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rituximab + PCI-32765 (Experimental): Rituximab (375 mg/m2) given intravenously (IV) on Day 1, Day 8, Day 15, and Day 22, then continued once every 4 weeks only on Days 1 during cycles 2 - 6. PCI-32765 started on Day 2 of cycle 1 at a dose of 420 mg (3 * 140-mg capsules) orally daily and will be continued daily.
  Interventions: Drug: Rituximab; Drug: PCI-32765

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 intravenously on Day 1, Day 8, Day 15, and Day 22, then continued once every 4 weeks only on Days 1 during cycles 2 - 6.
  Other Names: Rituxan
Drug: PCI-32765 — 420 mg (3 * 140-mg capsules) orally started on Day 2 of cycle 1 once daily and will be continued daily.

SUMMARY:
The goal of this clinical research study is to learn if PCI-32765 (Ibrutinib) combined with rituximab can help to control CLL and SLL. The safety of this combination will also be studied.

Ibrutinib is designed to stop a protein from working in the cells, which may cause the cancer cells to die or stop growing.

Rituximab is designed to attach to cancer cells and damage them, which may cause the cells to die.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive rituximab by vein on Days 1, 8, 15, and 22 of Cycle 1 (+ 3 days) and then on Day 1 (+/- 7 days) of Cycles 2-6.

Each cycle is 28 days.

You will take Ibrutinib capsules by mouth 1 time each day starting on Day 2 of Cycle 1. You should take it with 1 cup (8 ounces) of water.

You will also take allopurinol by mouth 1 time each day during the first 1-2 weeks of study treatment to lower the risk of side effects.

Study Visits:

On Days 7, 14, 21, and 28 of Cycle 1 (+/- 3 days):

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will be asked about any drugs you may be taking.

At the end of Cycles 2, 3, 4, 6, 9, and 12 (+/- 1 month):

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will be asked about any drugs you may be taking.

At the end of Cycles 3 or 6, and 12 (+/- 1 month), and then every 12 cycles (+/- 1 month) after that if the doctor thinks it is needed, you will have CT scans of the chest, abdomen and pelvis to check the status of the disease.

At the end of Cycles 3, 6, and 12 and then every 12 cycles (+/- 1 month) after that, you will have a bone marrow aspiration to check the status of the disease. If the doctor things these bone marrow aspirations are no longer needed, you will no longer have to have them.

Every 3 months (+/- 1 month) for Cycles 13-36 and every 6 months (+/- 1 month) after that:

* You will have a physical exam, including measurement of your vital signs.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will be asked about any drugs you may be taking.

Length of Treatment:

You may continue taking the study drug combination of rituximab and Ibrutinib for up to 6 cycles, after which Ibrutinib will be continued for up to a total of 12 cycles. It will be possible to continue with Ibrutinib treatment beyond 12 cycles if the study doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

This is an investigational study. Ibrutinib is FDA approved and commercially available for the treatment of patients with mantle cell lymphoma, CLL and SLL. Its use in this study is investigational. Rituximab is FDA approved to treat CLL and SLL.

Up to 40 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 1.Patients must have a diagnosis of high-risk CLL/SLL and be previously treated with up to 3 lines of prior therapy. High-risk CLL and high-risk SLL is defined by the presence of a 17p deletion or 11q deletion or TP53 mutation. Any CLL and SLL patient who has a short remission duration of less than 3 years after prior first-line chemo-immunotherapy, such as the FCR regimen, also fulfills criteria of high-risk CLL/SLL, regardless of the presence or absence of cytogenetic abnormalities.
2. 2.CLL and SLL patients with 17p deletion or TP53 mutation will not be required to have received any prior therapy, given the poor outcome of CLL/SLL patients to standard frontline chemo-immunotherapy, such patients will be eligible if they are untreated or if they have received up to 3 lines of prior therapy.
3. Patients must have an indication for treatment by 2008 IWCLL Criteria.
4. Patients age > 18 years at the time of signing informed consent. Understand and voluntarily sign an informed consent. Be able to comply with study procedures and follow-up examinations.
5. Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) performance status of 0-1.
6. Patients of childbearing potential must be willing to practice highly effective birth control (e.g., condoms, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], sexual abstinence, or sterilized partner) during the study and for 30 days after the last dose of study drug. Women of childbearing potential include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Post menopause is defined as follows: Amenorrhea >/= 12 consecutive months without another cause and a documented serum follicle stimulating hormone (FSH) level >35 mIU/mL; a male of childbearing potential is any male that has not been surgically sterilized.
7. Adequate renal and hepatic function as indicated by all of the following: Total bilirubin </=1.5 x institutional Upper Limit of Normal (ULN) except for patients with bilirubin elevation due to Gilbert's disease who will be allowed to participate; an Alanine (ALT) </=2.5 x ULN; and an estimated creatinine clearance (CrCl) of > 30 mL/min, as calculated by the Cockcroft-Gault equation unless disease related.
8. Free of prior malignancies for 3 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma in situ of the cervix or breast.
9. A Urine Pregnancy Test (within 7 days of Day 1) is required for women with childbearing potential

Exclusion Criteria:

1. Pregnant or breast-feeding females.
2. Treatment including chemotherapy, chemo-immunotherapy , monoclonal antibody therapy, radiotherapy, high-dose corticosteroid therapy (more than 60 mg prednisone or equivalent daily), or immunotherapy within 21 days prior to enrollment or concurrent with this trial.
3. Investigational agent received within 30 days prior to the first dose of study drug or have previously taken PCI-32765. If received any investigational agent prior to this time point, drug-related toxicities must have recovered to Grade 1 or less prior to first dose of study drug.
4. Systemic fungal, bacterial, viral, or other infection not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
5. Patients with uncontrolled Autoimmune Hemolytic Anemia (AIHA) or autoimmune thrombocytopenia (ITP).
6. Patients with severe hematopoietic insufficiency, as defined by an absolute neutrophil count of less than 500/micro-L and/or a platelet count of less than 30,000/micro-L at time of screening for this protocol.
7. Any other severe concurrent disease, or have a history of serious organ dysfunction or disease involving the heart, kidney, liver or other organ system that may place the patient at undue risk to undergo therapy with PCI-32765 and rituximab.
8. Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
9. Significant screening ECG abnormalities including left bundle branch block, 2nd degree AV block type II, 3rd degree block, bradycardia, and QTc > 470 msec.
10. Any serious medical condition, laboratory abnormality, or psychiatric illness that places the subject at unacceptable risk if he/she were to participate in the study.
11. History of stroke or cerebral hemorrhage within 6 months.
12. Evidence of bleeding diathesis or coagulopathy.
13. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 1, anticipation of need for major surgical procedure during the course of the study.
14. Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to Day 1. Bone marrow aspiration and/or biopsy are allowed.
15. Serious, non-healing wound, ulcer, or bone fracture.
16. Treatment with Coumadin. Patients who recently received Coumadin must be off Coumadin for at least 7 days prior to start of the study.
17. Any chemotherapy (e.g., bendamustine, cyclophosphamide, pentostatin, or fludarabine), immunotherapy (e.g., alemtuzumab, or ofatumumab), bone marrow transplant, experimental therapy, or radiotherapy is prohibited during therapy on this study.
18. Use of medications known to prolong QTc interval or that may be associated with Torsades de Pointes (refer to Appendix F) are prohibited within 7 days of starting study drug and during study-drug treatment.
19. Requires treatment with strong CYP3A4/5 and/or CYP2D6 inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-02-27 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan A. Burger, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Burger JA, Keating MJ, Wierda WG, Hartmann E, Hoellenriegel J, Rosin NY, de Weerdt I, Jeyakumar G, Ferrajoli A, Cardenas-Turanzas M, Lerner S, Jorgensen JL, Nogueras-Gonzalez GM, Zacharian G, Huang X, Kantarjian H, Garg N, Rosenwald A, O'Brien S. Safety and activity of ibrutinib plus rituximab for patients with high-risk chronic lymphocytic leukaemia: a single-arm, phase 2 study. Lancet Oncol. 2014 Sep;15(10):1090-9. doi: 10.1016/S1470-2045(14)70335-3. Epub 2014 Aug 20. PMID 25150798
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Details: February 2012 - September 2012
Period: Overall Study
Arm/Group | Rituximab + PCI-32765
Started | 40
Completed | 40
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab + PCI-32765
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 65 [35 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 37
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival defined as the time interval from treatment to progressive disease or death, whichever happens earlier. Participants in complete remission (CR), partial remission (PR) or stable disease (SD) are all counted as progression-free. Survival or times to progression functions estimated using the Kaplan-Meier method.
Time Frame: up to 50 months
Population: 1 participant was not evaluable for response
Measure: Median (Full Range); unit: Months
Arm/Group | Rituximab + PCI-32765
Number analyzed (Participants) | 39
Months | 45 [2 to 50]

2. Primary Outcome: Number of Participants With a Response
Description: Over all Response = complete remission (CR) + partial remission (PR). Complete remission (CR), requiring absence of peripheral blood clonal lymphocytes by immunophenotyping, absence of lymphadenopathy, absence of hepatomegaly or splenomegaly, absence of constitutional symptoms and satisfactory blood counts; positive or negative minimal residual disease (MRD); Partial remission (PR), defined as ≥ 50% fall in lymphocyte count, ≥ 50% reduction in lymphadenopathy or ≥ 50% reduction in liver or spleen, together with improvement in peripheral blood counts
Time Frame: 7 months
Population: 1 participant was not evaluable for response
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab + PCI-32765
Number analyzed (Participants) | 39
Participants | 37

ADVERSE EVENTS:
Time Frame: 7 months
Arm/Group | Rituximab + PCI-32765
All-Cause Mortality (participants affected / at risk) | 2/40
Serious Adverse Events (participants affected / at risk) | 18/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab + PCI-32765 (N=40)
Abdominal Pain (General disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (3)
Cardiac disorders - other (Cardiac disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Eye disorders - other (Eye disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Lung Infection (Infections and infestations) | 9 (11)
Mucosal infection (Infections and infestations) | 1 (1)
Musculoskeletal and connective tissue disorder - other (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1)
Renal and urinary disorders - other (Renal and urinary disorders) | 1 (3)
Respiratory, thoracic and mediastinal disorders - other (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Sepsis (Infections and infestations) | 3 (3)
Wound Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab + PCI-32765 (N=40)
Lung Infection (Infections and infestations) | 11 (11)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Diarrhea (Gastrointestinal disorders) | 10 (10)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fatigue (General disorders) | 7 (7)
Nausea/vomiting (Gastrointestinal disorders) | 15 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 (11)
Bleeding event (Blood and lymphatic system disorders) | 13 (13)
Peripheral Neuropathy (Nervous system disorders) | 3 (3)
Weight Gain (Investigations) | 4 (4)
Eye disorders (Eye disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (4)
Headache (General disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Hot flashes (Vascular disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-11-13): https://cdn.clinicaltrials.gov/large-docs/19/NCT01520519/Prot_SAP_000.pdf